CLINICAL TRIAL: NCT01784146
Title: Analysis of the Distribution of Pulmonary Ventilation After Nebulization by Heliox Associated With Positive Expiratory Pressure in Patients Asthmatics Stable.
Brief Title: Plethysmography Opto-electronic and Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Daniella Cunha Brandao, PhD, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Luciana 2
Record Dates: First submitted 2013-01-30; First posted 2013-02-05 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2012-12

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Oxygen; heliox

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Oxygen (Placebo Comparator)
  Interventions: Other: Oxygen
- PEEP + Heliox (Experimental)
  Interventions: Other: Heliox; Other: PEEP
- Oxygen + PEEP (Experimental)
  Interventions: Other: Oxygen; Other: PEEP
- Heliox (Active Comparator)
  Interventions: Other: Heliox

INTERVENTIONS:
Other: Oxygen — For inhalation of oxygen, we used a noninvasive delivery system, semi - closed (Figure 3) consisting of a non-toxic face mask with two unidirectional valves - inspiratory and expiratory branch - connected to the
  nebulizer (Airlife Misty Neb, Baxter; Valencia, CA, USA). In the inspiratory branch, a reservoir bag (Hudson RCI, USA) with capacity of 2.5 L was connected, in order to avoid dilution of the gas. This skin was fixed to the patient's face to prevent leakage and to maintain adequate pressurization and improved patient compliance to the PEEP. The nebulizer was fed by a flow of 8 l / min of oxygen.
  Arms: Oxygen; Oxygen + PEEP
Other: Heliox — For inhalation of heliox, we used a noninvasive delivery system, semi - closed consisting of a non-toxic face mask with two unidirectional valves - inspiratory and expiratory branch - connected to the
  nebulizer (Airlife Misty Neb, Baxter; Valencia, CA, USA). In the inspiratory branch, a reservoir bag (Hudson RCI, USA) with capacity of 2.5 L was connected, in order to avoid dilution of the gas. This skin was fixed to the patient's face to prevent leakage and to maintain adequate pressurization and improved patient compliance to the PEEP. The nebulizer was fed by a 11 l / min of heliox for the heliox group in accordance with a protocol of Hess et al.
  Arms: Heliox; PEEP + Heliox
Other: PEEP — PEEP supplied was 10 cm H2O through valve (Vital Signs,Totowa, USA) attached to the expiratory branch.
  Arms: Oxygen + PEEP; PEEP + Heliox

SUMMARY:
Objective: To assess the influence of nebulization with bronchodilators carried by the heliox coupled to PEP in the distribution of compartimental lung volumes in asmathic adults and to correlate with pulmonary function data. Methods: A controlled randomized trial involving 27 patients divided into four groups: heliox + PEP, oxygen + PEP, heliox and oxygen. After the initial evaluation, it was placing 89 reflective markers attached to the surface of the trunk and images acquired by optoelectronic plethysmography (OEP) of six cameras. Three slow vital capacity maneuvers and quiet breathing regarded as phase control. After the control phase, all patients underwent nebulization with a distribution noninvasive system, semi-closed using 10 drops of Fenoterol Bromide and 20 drops of Ipratropium.

ELIGIBILITY:
Inclusion Criteria:

* The study included individuals diagnosed with moderate to severe asthma with forced expiratory volume in one second (FEV1) <60% or FEV1 <60% - 80% predicted;
* showing reversibility of bronchial obstruction after administration of bronchodilators at least 10% in FEV1.

Exclusion Criteria:

* unable to understand or perform the spirometric maneuver;
* with a history of smoking;
* pulmonary comorbidities as chronic obstructive pulmonary disease (COPD);
* bronchiectasis and tuberculosis sequel;
* hemodynamic instability defined as heart rate (HR) greater than 150 bpm or systolic blood pressure below 90 mmHg or greater than 150mmHg;
* pregnancy and any contraindication to the use of PEEP;
* such as increased work of breathing (acute asthma);
* active hemoptysis;
* acute sinusitis;
* pneumothorax;
* untreated; surgery or facial trauma;
* oral or injury;
* epistaxis;
* nausea and esophageal surgery.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2009-06; Primary Completion 2009-06 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Distribution of volumes of the rib cage in asthma patients-Plesthysmography opto - electronic (POE). | 5 months
  The markers are meant to reflect the infrared signal emitted by the POE to the sensors, which transform these signals into information about the movement of the chest. In this evaluation method the chest is considered a geometric model divided into three regions - the volume of pulmonary rib cage (Vrp), abdominal rib cage volume (Vra), part of the chest corresponding to the diaphragm, and abdomen (Va), and the overall volume of the chest (Vcw) the total volume of compartments.

SECONDARY OUTCOMES:
Lung function in asthmatic subjects | 5 mothns
  In spirometry values were obtained for FEV1, PEF and forced vital capacity (FVC), considering the record as the best value according to the American Thoracic Society 18 the percentage of the predicted 16. For IC, we performed a correction of the weight. The present study included all patients were instructed to discontinue their medication twelve hours before the experiment as corticosteroids and bronchodilators for short or long duration for performing spirometry

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratório de Fisiologia e Fisioterapia cardiorespiratória, Recife, Pernambuco, Brazil

REFERENCES:
- [Result] Frischknecht-Christensen E, Norregaard O, Dahl R. Treatment of bronchial asthma with terbutaline inhaled by conespacer combined with positive expiratory pressure mask. Chest. 1991 Aug;100(2):317-21. doi: 10.1378/chest.100.2.317. PMID 1864100
- [Result] Manthous CA, Hall JB, Caputo MA, Walter J, Klocksieben JM, Schmidt GA, Wood LD. Heliox improves pulsus paradoxus and peak expiratory flow in nonintubated patients with severe asthma. Am J Respir Crit Care Med. 1995 Feb;151(2 Pt 1):310-4. doi: 10.1164/ajrccm.151.2.7842183.